CLINICAL TRIAL: NCT05413473
Title: Northern Alberta Linac-MR Image-Guided Human Clinical Trials - 2
Brief Title: Northern Alberta Linac-MR Image-Guided Radiotherapy (Northern LIGHTs-2)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-0019
Record Dates: First submitted 2022-06-03; First posted 2022-06-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MR guided radiotherapy (Experimental): MR-guided radiotherapy using the Alberta linac-MR P3 system. Contemporary radiotherapy techniques and fractionation schedules will be conducted in the following graduated stages with overlap between stages allowed:
  Stage 1: Parallel-opposed pair treatments (palliative) Stage 2: 4 field box treatments (curative or palliative) Stage 3: High dose treatments - multi-field 3DCRT (curative or palliative) Stage 4: High dose treatments - multi-field IMRT (curative or palliative)
  Interventions: Device: MR guided radiotherapy

INTERVENTIONS:
Device: MR guided radiotherapy — MR guided radiotherapy using the Alberta linac-MR P3 system
  Other Names: Alberta linac-MR P3 system

SUMMARY:
Cancers are often treated with external beam radiotherapy. Current radiotherapy treatments are performed using computed tomography (also known as CT) scans which may not always clearly identify the cancer. In some instances, magnetic resonance imaging (MRI) may be able to better identify cancers. Therefore, efforts are currently underway to use the MRI scans to improve radiotherapy treatments or eventually even use radiotherapy equipment that only uses MRI scans to guide treatments. This new technology that will only use MRI scans to guide treatments is called the Linac-MR (linear accelerator with an MRI). This new Linac-MR is a unique innovation at the Cross Cancer Institute, with theoretical advantages over other Linac-MR machines that are being tested elsewhere in the world. This feasibility study is being done as a first step in clinical development of the Linac-MR, as this new technology has to be tested to see if it is acceptable to both doctors and participants. The purpose of this Phase I/II study is (1) to verify treatment completion as intended and scheduled the oncology team, and (2) to evaluate treatment effects, including any expected or unexpected radiation side effects and cancer response to radiation. This study will allow the researchers at the Cross Cancer Institute to develop this technology further by conducting additional studies to take advantage of MRI scanning on tumor tracking during radiation treatments.

DETAILED DESCRIPTION:
This prospective, open-label, Phase I/II, clinical trial is feasibility study to evaluate MR-guided radiotherapy with the Alberta linac-MR P3 system in adult patients with cancer that are treated with external beam radiotherapy in four graduated stages (described below), progressing from palliative participants with simple techniques to curative participants with complex techniques, with progression to each stage determined by an internal SAFE review committee. Conventional treatment margins and doses will be utilized, with the MR being utilized in place of CT based imaging. The intent is to replicate current CT based treatments on the Alberta linac-MR P3 system using MR guided imaging, planning and treatment delivery. MR imaging will be utilized for simulation, planning and image guidance. Dosimetry will be done as per standard of care. MRI contrast may be used, as applicable. Adverse events will be collected weekly during RT, and participants will complete one questionnaire at the end of their RT treatment. Follow-up will consist of adverse event assessment at 1, 6, and 12 months following completion of RT, and may be assessed annually via chart review for up to 1 year. Survival status will be assessed at 12 months following completion of RT, and then annually for up to 1 year.

In stage 1, 4 to 15 participants with incurable malignancies that require palliative radiotherapy with parallel-opposed pair beam arrangements will be enrolled. These will be patients with bone or brain metastases from their malignancies that require either a single fraction or multiple fractions of radiotherapy. The treatment will be a simple opposed pair beam arrangement to a dose of a single 8 Gy or to a dose of 20 Gy over a course of 5 fractions. Once some initial treatments are completed, and at the discretion of an internal SAFE review committee, additional treatment sites will be permitted (i.e. lung, abdomen, etc.) that are also utilizing a simple opposed pair beam arrangement with the above doses.

In stage 2, 10 to 28 participants with malignancies (curative or palliative treatments) that require multi-field arrangement for their external beam radiotherapy will be enrolled. Initially, 4 field techniques (anterior, posterior, right lateral, left lateral) will be utilized to treat central tumors using fractionation schemes that are currently considered standard of care. Patients with pelvic malignancies (i.e. prostate cancers, rectal cancers, cervical cancers, endometrial cancers) or other malignancies requiring simple four field techniques will be identified for this stage.

In stage 3, 5 to 28 participants with malignancies (curative or palliative) that require more complicated multi-field 3DCRT treatments (not requiring IMRT) to a high radiation dose for their external beam radiotherapy (i.e. lung, brain, etc.) will be enrolled. This will include the use of field-in-field techniques such as step-and-shoot techniques to allow for modulation of the radiation beam during treatment.

In stage 4, 10 to 28 participants with malignancies (curative or palliative) that require more complicated multi-field IMRT treatments for their external beam radiotherapy (i.e. prostate, head and neck, lung, brain, etc.) will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Patients deemed fit to undergo external beam radiation therapy by their attending radiation oncologist
* Accessible for follow-up

Exclusion Criteria:

* Patients with contraindications for MRI
* Patients who are unable to lie flat and still for the duration of the expected scan acquisition and treatment
* Patients who are unable to provide informed consent
* Patients with clinically significant inferior treatment plans compared to standard CT based external beam plans. For example, plans that generate hot spots of > 110% or other unacceptable treatment plans that would not otherwise arise with standard CT based external beam plans.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of planned radiotherapy fractions that are administered, without clinically unacceptable interruptions, with the Alberta linac-MR P3 system. | Approximately 6 years
  The total number of planned radiotherapy fractions that are administered, without clinically unacceptable interruptions, on the Alberta linac-MR P3 system. The study will track the number of planned fractions administered per participant without any significant interruptions or delays in their treatment.

SECONDARY OUTCOMES:
Incidence of acute toxicity | 6 months post treatment
  Acute toxicity (within 6 months post treatment) graded according to CTCAE version 5.0 will be assessed when all participants have completed a minimum of 1 year follow-up.
Incidence of late toxicity | between 6 months and 2 years post treatment
  Late toxicity (greater than 6 months post treatment) graded according to CTCAE version 5.0 will be assessed when all participants have completed a minimum of 1 year follow-up.
Quantify the patient experience on the Linac-MR | 1 year post treatment
  Participants will complete a questionnaire at the end of their MR guided radiotherapy. The questionnaire will assess participant comfort and their perception of the treatment experience using a 1 - 5 scale.
Overall treatment time | 1 year post treatment
  The total MR guided radiotherapy time will be recorded for each participant, which is comprised of the sum of time the participant is in the treatment room and the total treatment time daily. The overall treatment duration should not exceed the original scheduled treatment duration via conventional radiotherapy by more than five business days, in case of unexpected servicing needs or any other delays.
Overall treatment planning time | 1 year post treatment
  The total treatment planning time using the Linac-MR will be recorded for each participant. The overall treatment planning time should be within the currently accepted ready to treat timelines for conventional radiotherapy.
Time to local control | Up to 2 years after completion of treatment
  Time from treatment until the recurrence of disease locally.
Disease-free survival | Up to 2 years after completion of treatment
  Time from treatment until the recurrence of disease (or death).
Overall survival | Up to 2 years after completion of treatment
  Time from treatment until death from any cause. Survival status will be assessed at 12 months following completion of treatment, then annually for up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Nawaid Usmani, MD, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No